

Doküman Kodu: ÜNV-KAEK-DYD-005

Yayın Tarihi: 30.03.2022

Revizvon No: 01

Revizyon Tarihi: 01.06.2022

Sayfa 1 / 5

#### STUDY PROTOCOL

1. Date: 01.01.2023

#### 2. Official Title:

THE EFFECT OF A NEWLY FORMULATED PREOPERATIVE ORAL CARBONHYDRATE SOLUTION ON GASTRIC EMPTYING, POSTOPERATIVE NAUSEA AND VOMITING AND STRESS RESPONSE

#### 3. **Method:**

109 patients who underwent elective laparoscopic cholecystectomy, aged 18-65 years and ASA physical state 1-2 were included in the study. The patients were divided into 3 groups: Group A, who would not eat anything 6-8 hours before the operation, Group S, who drank 400 ml of water 2 hours before the operation, and Group K, which drank 400 ml preoperative oral carbohydrate solution (PreOKH) 2 hours before the operation. Before induction of anesthesia (T1), patients antral gastric cross-sectional area (GKA) and gastric volume (GV) were evaluated by gastric ultrasound. The preoperative anxiety level of the patients was determined by the State-Trait Anxiety Inventory (STAI) before the operation (T1), and the symptoms affecting the preoperative patient comfort parameters (thirst, hunger, dry mouth, fatigue) were measured 2 hours before the operation (T0) and before the induction (T1) evaluated with the visual analog scale (VAS). Postoperative nausea and vomiting (PONV) and postoperative pain levels were recorded. Blood glucose, insulin and cortisol levels of the patients were measured 2 hours before the operation (T0), before induction (T1) and postoperative 2nd hour (T3).

Descriptive statistics of qualitative variables in the study will be given as number and percentage, and descriptive statistics of quantitative variables will be given as mean, median, standard deviation, minimum and maximum. Pearson chi-square and Fisher's exact chi-square tests will be used to compare the distribution of the relevant variables between the groups. The conformity of quantitative variables to normal distribution will be examined by Shapiro Wilk test. For normally distributed variables, one-way analysis of variance will be used to compare the means of more than two groups. Tukey test will be used as a posthoc test for pairwise comparisons. For non-normally distributed variables, Kruskall Wallis test will be used in the mean comparison of more than two groups and pairwise comparisons will be examined with Dunn test. Paired t test will be used for the mean comparison of two dependent groups and Wilcoxon signed-rank test will be used for median comparisons. Repeated measures analysis of variance method will be used for mean comparisons of more than two dependent groups and Friedman test will be used for median comparisons. Statistical significance level will be taken as 0.05 and SPSS (Version 28) package program will be used for calculations. For the gastric volume value, at the 95% confidence level, when the significance of a mean difference of 18.18 with 80% power is attributed (means 67.22 and 49.04 with standard deviations 29.49 and 15.4), a minimum of 28 people should be included in the study in each group. [1] Therefore, we planned the number of patients in the study groups as 30 for each group. 1



Doküman Kodu: ÜNV-KAEK-DYD-005

Yavın Tarihi: 30.03.2022

Revizyon No: 01

Revizyon Tarihi: 01.06.2022

Sayfa 2 / 5

#### **Inclusion Criteria:**

- 1. Between the ages of 18-65
- 2. Elective laparoscopic cholecystectomy planned under general anesthesia
- 3. American Society of Anesthesiologists (ASA) class I-II physical condition

### **Exclusion Criteria:**

- 1. Patients with gastroesophageal reflux and gastrointestinal motility disorders
- 2. diabetes mellitus
- 3. Mental retardation, previous neurological disease symptoms (syncope, dementia, alzheimer etc.)
- 4. Chronic alcoholism
- 5. Difficult Intubation
- 6. Patients with ASA physical status classes ≥III
- 7. Patients with a body mass index of 35 and above
- 8. History of meniere and motion sickness
- 9. Presence of previous history of postoperative nausea and vomiting
- 10. Smoking

### Numerik Rank Score:

0: no vomiting or nausea

1: nausea

2:nausea and once vomiting

3:twice or more vomiting

## VAS:



### Qualitative evaluation of the antrum with gastric USG:

Grade 0: empty antrum both in the semi-sitting position and in the RLDP

Grade 1: gastric fluid is only visible in RLDP;

Grade 2: gastric fluid can be seen both in the semi-sitting position and in RLDP



Doküman Kodu: ÜNV-KAEK-DYD-005

Yayın Tarihi: 30.03.2022

Revizyon No: 01

Revizyon Tarihi: 01.06.2022

Sayfa 3 / 5

# Factor Loading

| Item | Ī | II | h <sup>2</sup> |
|---|---|---|---|
| 1. I feel calm | .50 | 21 | .41 |
| 2. I feel secure | .61 | 10 | .45 |
| 3. I am tense | .01 | .63 | .39 |
| 4. I am strained | .05 | .59 | .32 |
| 5. 1 feel at ease | .59 | 05 | .38 |
| 6. I feel upset | .03 | .78 | .58 |
| 7. I am presently worrying | 01 | .57 | .33 |
| 8. I feel satisfied | .57 | 10 | .39 |
| 9. I feel frightened | 03 | .69 | .50 |
| 10. I feel comfortable | .59 | 19 | .51 |
| 11. I feel self-confident | .70 | .04 | .46 |
| 12. I feel nervous | .05 | .76 | .54 |
| 13. I feel jittery | .01 | .73 | .52 |
| 14. I feel indecisive | 09 | .55 | .37 |
| 15. I am relaxed | .58 | -,10 | .41 |
| 16. I feel content | .62 | .06 | .35 |
| 17. I am worried | .12 | .79 | .54 |
| 18. I feel confused | 10 | .62 | .45 |
| 19. I feel steady | .69 | 01 | .47 |
| 20. I feel pleasant | .68 | .05 | .43 |
| 21. I feel pleasant | .64 | .02 | .40 |
| 22. I tire nervous and restless | 32 | .44 | .44 |
| 23. I feel satisfied with myself | .79 | .09 | .5€ |
| 24. I wish I could be as happy as others seem | 20 | .23 | .14 |
| 25. I feel like a failure | 48 | .15 | .32 |
| 26. I feel rested | .61 | .09 | .33 |
| 27. I am calm, cool, and collected | .67 | .03 | .43 |
| 28. I feel that difficulties are piling | 34 | .38 | .39 |
| 29. I worry too much over something | 06 | .37 | .1€ |
| 30. I am happy | .70 | 05 | .52 |
| 31. I am inclined to take things hard | 20 | .38 | .27 |
| 32. I lack self-confidence | 38 | .17 | .25 |
| 33. I have disturbing thoughts | .78 | .03 | .59 |
| 34. I make decisions easily | .50 | .02 | .27 |
| 35. I feel inadequate | 38 | .21 | .27 |
| 36. I am content | .70 | 07 | .55 |
| 37. Some unimportant thought runs | 10 | .34 | .16 |
| 38. I take disappointments so keenly | 26 | .28 | .22 |
| 39. I am a steady person | .52 | 08 | .32 |
| 40. I get in a state of tension or turmoil | 38 | .30 | .35 |

Note. Interfactor correlation = -0.52. Factor loadings are standardized regression coeff



Doküman Kodu: ÜNV-KAEK-DYD-005

Yayın Tarihi: 30.03.2022

Revizyon No: 01

Revizyon Tarihi: 01.06.2022

Sayfa 4 / 5

## **FOLLOW-UP FORM**

| No: | Duration of operation | |
|------------|------------------------------|---------------|
| Age-gender | Fasting time | |
| BMI | Anesthetic agent consumption | Sevoflurane: |
| GRUP | | Remifentanil: |
| ASA | complications: | |
| disease | Antiemetic need : | |

## **Gastric examination**

| Gastrik USG – measurement of CSA in RLPD | LD: | SD: | CSA: |
|---|---|---|---|
| $(CSA = (LD \times SD \times \pi)/4)$ | | | |
| Gastric volume | | | |
| $(GV = 27.0 + 14.6 \times CSA (RLDP'de) - 1.28 \times age)$ | | | |
| Qualitative evaluation score | | | |
| Gastiric volume (aspiration of ngs) | | | |
| Gastric pH | | | |

# **Intraoperative vital sing**

| | HR | SP/DP | MAP | SpO <sub>2</sub> | BİS |
|-------------------|----|-------|-----|------------------|-----|
| Before induction | | | | | |
| İnd +1. min | | | | | |
| 10.min | | | | | |
| 20. min | | | | | |
| 30. min | | | | | |
| 40. min | | | | | |
| 50. min | | | | | |
| 60. min | | | | | |
| Before extubation | | | | | |
| After extubation | | | | | |



Doküman Kodu: ÜNV-KAEK-DYD-005 Yayın Tarihi: 30.03.2022 Revizyon No: 01 Revizyon Tarihi: 01.06.2022 Sayfa 5 / 5

| PACU 1. min |
|-------------|
| PACU 15.min |

| | STAI | VAS | PONK | Glucose | Insulin | cortisole |
|------------------|------|-----|------|---------|---------|-----------|
| Preop 2. hours | | | | | | |
| Berofe induction | | | | | | |
| PACU | | | | | | |
| Postop 2. hours | | | | | | |
| Postop 12. hours | | | | | | |
| discharge | | | | | | |

Koordinatör: Prof. Dr. Kazım Karaaslan

İmza

## References

1) Zhang Z, Wang RK, Duan B, Cheng ZG, Wang E, Guo QL, Luo H. Effects of a Preoperative Carbohydrate-Rich Drink Before Ambulatory Surgery: A Randomized Controlled, Double-Blinded Study. Med Sci Monit. 2020 Aug 28;26:e922837. doi: 10.12659/MSM.922837